CLINICAL TRIAL: NCT05561231
Title: A Prospective Single Blinded Randomised Controlled Trial to Compare Endotracheal Intubation Using C Blade and D Blade of CMAC Videolaryngoscope in Patients Undergoing Elective Cervical Spine Surgery
Brief Title: Comparing Ease of Endotracheal Intubation Using C Blade and D Blade of CMAC Videolaryngoscope in Patients Undergoing Elective Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Memorial Hospital, Mumbai (Other Government)
Responsible Party: Principal Investigator, Sandhya Narayanan P, Principle investigator, King Edward Memorial Hospital, Mumbai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EC/182/2018
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Cervical Spine Instability
Keywords: Manual in-line stabilisation; C blade; D blade
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Intervention Model Description: Prospective single blinded randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Active Comparator): Group of patients intubated with C blade of CMAC videolaryngoscopes
  Interventions: Procedure: Intubation with C blade
- Group D (Active Comparator): Group of patients intubated with D blade of CMAC videolaryngoscope
  Interventions: Procedure: Intubation with D blade

INTERVENTIONS:
Procedure: Intubation with C blade — Intubation with C blade of CMAC videolaryngoscope
  Arms: Group C
Procedure: Intubation with D blade — Intubation with D blade of CMAC videolaryngoscope
  Arms: Group D

SUMMARY:
This study was done to compare the ease of tracheal intubation using the conventional C blade and the D blade of CMAC videolaryngoscope in patients undergoing cervical spine surgery.

DETAILED DESCRIPTION:
Manual in-line stabilisation is used to immobilise the neck during endotracheal intubation in patients undergoing cervical spine surgery to prevent secondary spinal cord damage. This makes visualisation of the glottis difficult with conventional laryngoscopy which can be overcome with videolaryngoscope. CMAC Videolaryngoscope has the conventional blade (C blade) and the highly angulated D blade which was introduced to aid in difficult airway. This study was done to compare the ease of tracheal intubation using the conventional C blade and the D blade of CMAC videolaryngoscope in patients undergoing cervical spine surgery.

Methodology: After Institutional Ethics Committee approval and obtaining informed consent, 68 patients undergoing elective cervical spine surgery were randomised into 2 groups - C (intubated with C blade) or D (intubated with D blade) (n=34 each) by computer generated randomisation. After induction of general anaesthesia, manual in-line stabilisation of the cervical spine was achieved and intubation was attempted by experienced anaesthesiologist with the C blade or D blade according to the group. The time taken for successful intubation, time taken for optimum glottic visualisation, the number of attempts, additional manouvres required for successful intubation and the incidence of complications were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA (American Society of Anaesthesiology) grade one and two,
* aged 18 years and older,
* Patients with mouth opening more than two and a half fingers (inter-incisor distance >3cm)

Exclusion Criteria:

* Patients who were unwilling to be a part of the study,
* patients with any oral pathology, hiatus hernia, pregnant women,
* patients with severe systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Time taken for successful intubation | During procedure
  Comparing the time taken for successful intubation using the C blade and D blade of CMAC videolaryngoscope in patients with manual in-line stabilisation of the cervical spine

SECONDARY OUTCOMES:
Time taken to obtain the best Cormack-Lehane grade | During procedure
  Comparing the time taken to obtain the best Cormack-Lehane grade using the C blade and D blade of CMAC videolaryngoscope in patients with manual in-line stabilisation of the cervical spine
Number of attempts, external manouvres, complications | During procedure
  Comparing the number of attempts for successful endotracheal intubation, external manoeuvres or adjuncts required, complications caused using the C blade and D blade of CMAC videolaryngoscope in patients with manual in-line stabilisation of the cervical spine

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya N Narayanan P, MD, Principal Investigator — Seth GSMC and KEMH Mumbai
Locations (1):
- Seth GSMC and KEM Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hazarika H, Saxena A, Meshram P, Kumar Bhargava A. A randomized controlled trial comparing C Mac D Blade and Macintosh laryngoscope for nasotracheal intubation in patients undergoing surgeries for head and neck cancer. Saudi J Anaesth. 2018 Jan-Mar;12(1):35-41. doi: 10.4103/sja.SJA_239_17. PMID 29416454
- [Background] Sinha R, Ray BR, Sharma A, Pandey RK, Punj J, Darlong V, Trikha A. Comparison of the C-MAC video laryngoscope size 2 Macintosh blade with size 2 C-MAC D-Blade for laryngoscopy and endotracheal intubation in children with simulated cervical spine injury: A prospective randomized crossover study. J Anaesthesiol Clin Pharmacol. 2019 Oct-Dec;35(4):509-514. doi: 10.4103/joacp.JOACP_106_18. PMID 31920236